CLINICAL TRIAL: NCT06577506
Title: Improving Access to Diabetes Education and Care for Deaf Populations
Brief Title: Diabetes Education and Care for Deaf Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Michelle Litchman, Principal Investigator, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00151575
Record Dates: First submitted 2023-11-07; First posted 2024-08-29 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Deaf Diabetes Can Together (Experimental)
  Interventions: Behavioral: Deaf Diabetes Can Together

INTERVENTIONS:
Behavioral: Deaf Diabetes Can Together — 10-week diabetes self-management telehealth intervention for deaf adults with diabetes.

SUMMARY:
This study will assess the feasibility and preliminary efficacy of a 10-week intervention called "Deaf Diabetes Can Together".

ELIGIBILITY:
Inclusion Criteria:

* Identify as Deaf/Hard of Hearing
* living with diabetes (any type)
* speak and understand English or American Sign Language
* have access to internet
* willing to participate in the intervention

Exclusion Criteria:

* participating in another diabetes study
* have significant cognitive impairment
* are pregnant or planning to become pregnant in the next year
* have life expectancy of <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
A1C Level | 6 months: (Test at 0 weeks, 12 weeks, and 24 weeks)
  Clinical outcome

SECONDARY OUTCOMES:
Diabetes Distress Level Using the Screening Scale Questionnaire | 6 months: (Test at 0 weeks, 12 weeks, and 24 weeks)
  Psychosocial outcome, scoring averaged from 1-6 with higher score means worse outcome.
Diabetes Self-Care Level using the Self-Care Inventory Revised Questionnaire | 6 months: (Test at 0 weeks, 12 weeks, and 24 weeks)
  Self-management outcome, scoring averaged from 0-100 point scale with higher score means better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided